CLINICAL TRIAL: NCT00752193
Title: Safety and Efficacy of a Vaginally Administered Probiotic Lactobacilli Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2008/438
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Probiotic lactobacilli
  Interventions: Other: Probiotic lactobacilli
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic lactobacilli — Probiotic lactobacilli in combination with antibiotic therapy
  Arms: 1
Other: Placebo — Placebo in combination with antibiotic therapy
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety and the efficacy of vaginally administered probiotic lactobacilli in combination with antibiotic therapy (metronidazole) in women with microbiologically defined bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Untreated Bacterial Vaginosis (BV) (asymptomatic or symptomatic) as diagnosed during the screening visit using Amsel criteria.
* Otherwise healthy? pre-menopausal women between 18-50 years of age at date of screening.
* Regular menstrual cycles (21-35 days) or amenorrheic for at least 3 months due to use of a long acting progestin or continuous use of oral contraceptives.
* Subject is willing to insert vaginal applicators.
* Subject is willing to be asked questions about personal medical health and sexual history
* Normal Pap smear collected at the screening visit? If a subject's Visit 0 Pap smear result is any of the following, the person is ineligible for participation: ASC-US (atypical squamous cells of undetermined significance), AGC (atypical glandular cells), ASC-H (atypical squamous cells, cannot r/o high grade lesion), LSIL (low grade squamous intraepithelial lesions), HSIL (high grade squamous intraepithelial lesions), adenocarcinoma in situ, adenocarcinoma, squamous cell carcinoma in situ, squamous cell carcinoma or inadequate sample
* Agree to be sexually abstinent 48 hours prior to Visit 1 (enrollment) until 48 hours after application of the study product and a second time after visit 2.
* Agree to abstain from the use of any other intravaginal product (i.e., contraceptive creams, gels, foams, sponges, lubricants, douches, etc.) throughout the trial period.
* Agree to use an adequate method of birth control for the duration of the study to avoid pregnancy. Acceptable methods include a history of tubal ligation, male partner with a vasectomy, a steroidal contraceptive (oral, patch, injectable or implantable), IUD (Paragard or Mirena), condoms or abstinence.
* Subject must have access to functioning refrigerator.

Exclusion Criteria:

* Urogenital infection at screening or within the 21 days prior to screening. This includes urinary tract infection, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis or Treponema pallidum. Subjects may be re-screened at least 21 days after the respective antibiotic or antifungal therapies have been completed.
* History of recurrent genital herpes.
* Diagnosis of N. gonorrhoeae, C. trachomatis, T. pallidum or T. vaginalis on two or more occasions during the six months prior to screening.
* Pregnancy or within 2 months of last pregnancy (all subjects will have a urine pregnancy test prior to enrollment).
* Lactation.
* Vaginal or systemic antibiotic or antifungal therapy within 21 days of the Screening visit or within 4 months of Enrollment visit.
* Investigational drug use within 4 months or 10 half-lives of the drug, whichever is longer, of enrollment visit. Planned investigational drug use while participating in this study.
* Menopause.
* IUD insertion or removal within the last 3 months.
* Pelvic surgery within the last 3 months.
* Cervical cryotherapy or cervical laser within the last 3 months.
* Use of a NuvaRing® within 3 days of the screening visit or during the course of the study.
* New long-acting treatments (e.g. depot formulation including medroxyprogesterone acetate (DMPA) form of hormonal birth control). Subjects may be enrolled if stable (> 3 months) on existing therapy as determined by the Principal Investigator.
* Diabetes or other significant disease or acute illness that in the Investigator's assessment could complicate the evaluation.
* Known HIV infection or positive HIV test at screening.
* Immunosuppressive drug within 4 months.
* Previous participation in a L. crispatus clinical study.
* Colposcopic findings at the enrollment visit involving significant deep disruption of the epithelium.
* Known allergy to any component (skim milk,…) of the drug or to latex (condoms).
* Unavailable for follow-up visits.
* History of drug or alcohol abuse.
* At enrollment, have any social or medical condition, or psychiatric illness that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The proposed research project aims at the development of a vaginal probiotic delivery system to restore and to maintain the vaginal microflora | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Temmerman, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be